CLINICAL TRIAL: NCT02747563
Title: Evaluation of PSA Blood Levels in Men on Active Surveillance and Men With Benign Prostatic Hyperplasia Prior to and After Digital Rectal Examination
Brief Title: Evaluation of PSA Blood Levels Prior to and After Digital Rectal Examination
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Dr Uri Lindner, Dr. Uri Lindner, Staff Urologist, Kaplan Medical Center, Kaplan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0210-15-KMC
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PSA; digital rectal examination
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Surveillance (Experimental): Patients with known prostate cancer eligible for active surveillance Intervention - PSA measurement
  Interventions: Other: Blood test (PSA)
- Controls (Active Comparator): Patients without known diagnosis of prostate cancer Intervention - PSA measurement
  Interventions: Other: Blood test (PSA)

INTERVENTIONS:
Other: Blood test (PSA) — Measurement of blood PSA levels

SUMMARY:
Patients with know prostate cancer (PCa) under active surveillance and aged matched controls without evidence of PCa will have a PSA blood test prior to and following standardized digital rectal examination

DETAILED DESCRIPTION:
Patients with know prostate cancer (PCa) under active surveillance (Gleason 6, PSA < 10 ng/ml) and aged matched controls without evidence of PCa will have a PSA blood test prior to and following standardized digital rectal examination.

The change of PSA will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Intact Rectum
* Prostate Cancer eligible for active surveillance

Exclusion Criteria:

* Pror radiation therapy
* Under Androgen Deprivation Therapy
* Prior prostate surgery

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of PSA elevation after DRE | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No